CLINICAL TRIAL: NCT07157293
Title: An Online Intervention To Enhance Motivation and Goal-Directed Behavior
Brief Title: Online Intervention To Improve Motivation
Acronym: Online Mot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lauren Luther, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300015163; Internal Award (Other Grant/Funding Number: University of Alabama at Birmingham)
Record Dates: First submitted 2025-08-25; First posted 2025-09-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia Prodromal; SCHIZOPHRENIA 1 (Disorder); Psychosis
Keywords: negative symptoms; schizophrenia; psychosis; digital health
MeSH Terms: conditions — Schizotypal Personality Disorder; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Motivation Focused Intervention (Experimental)
  Interventions: Behavioral: Online Motivation Enhancing Intervention

INTERVENTIONS:
Behavioral: Online Motivation Enhancing Intervention — This is a online intervention that will ask participants to review and complete 30 minutes of material each week.

SUMMARY:
Participants will complete one online intervention lasting 12 weeks. Each week, they will be asked to complete a 20-30 minute session online. The intervention is targeting improved mood and positive affect in order to support increases in motivation and goal-directed behavior. Before and after the intervention, participants will be asked to complete measures to assess symptoms, mood, and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or a related psychotic disorder
* Meeting criteria for being at clinical high risk for psychosis

Exclusion Criteria:

* Does not have access to a computer each week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Brief Negative Symptom Scale | immediately before and after the intervention
  Interview measure of motivation and pleasure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No